CLINICAL TRIAL: NCT06134518
Title: Effectiveness of the Education Program on Increasing the Competency Level of Health Cadres in Indonesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, Dewie Sulistyorini, Principal Investigator, Hiroshima University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 550/EA/KEPK-FKM/2023
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Maternal Mortality
Keywords: competency level, health cadre, maternal mortality
MeSH Terms: conditions — Maternal Death

STUDY DESIGN:
Intervention Model Description: Intervention group control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): The intervention group will receive the competency-based education program for 1 month at each PHC, after baseline data collection. The education program will be conducted weekly. This education session will be conducted for 4 hours per session, with 20 health cadres in a group per PHC .The competency level is measured by the researcher developing a competency questionnaire which consists of a knowledge test, skill, and attitude checklist score at the 2nd post-assessment (2 months after being given the education program).
  Interventions: Other: The education program
- control (Experimental): Health cadres in the control group have received the initial orientation from the PHCs. In this study, they take only the competency questionnaires including skill check will be collected following the data collection timeline. After completing the research, the control group will receive the education program material used for the intervention group if they require.
  Interventions: Other: the initial orientation from the PHCs

INTERVENTIONS:
Other: The education program — The intervention group will receive the competency-based education program for 1 month at each PHC, after baseline data collection. The education program will be conducted weekly. This education session will be conducted for 4 hours per session, with 20 health cadres in a group per PHC. The competency level is measured by the researcher developing a competency questionnaire which consists of a knowledge test, skill, and attitude checklist score at the 2nd post-assessment (2 months after being given the education program).
  Arms: intervention
Other: the initial orientation from the PHCs — the initial orientation from the PHCs
  Arms: control

SUMMARY:
Ending preventable maternal mortality (EPMM): By 2030, every country should reduce its maternal mortality ratio (MMR) by at least two-thirds from the 2010 baseline. In the era of the SDGs, an acceleration of current progress is required to achieve SGD target 3.1, working towards a vision of ending all preventable maternal mortality. In Central Java, one of the most effective efforts to reduce maternal mortality is increasing the number of human resources, who can assist pregnant mothers and supervise their period of pregnancy. The maternal mortality rate (MMR) in Banjarnegara Regency in 2021 is 287.05 per 100,000 live births, this indicates the top 10 in Central Java Province over the past 5 years. Health cadres, who are non-professional volunteer health supporters for pregnant women appointed by regional public health centers (PHCs), are expected to be the key human resources who contribute to reducing MMR in Indonesia and Banjarnegara Regency as well. However, based on an initial study by researchers conducting qualitative research with focus group discussions (FGDs) and in-depth interviews in April-July 2023, researchers found that health cadres had incorrect and unscientific knowledge. Therefore, improving the knowledge and skills of the health cadres through education programs could be expected to further improve the health outcomes of pregnant women, consequently contributing to reducing the MMR.

The purpose of this study is to improve health cadres' competency level in monitoring the risks of pregnant women. This monitoring activities for pregnant women by cadres is an effort to prevent maternal mortality, because if there are complications they can be treated as early as possible.

DETAILED DESCRIPTION:
1. Prior to the commencement of the study, the PI will visit the selected PHCs as the intervention group and control group, and then explain an overview of this study. The PI obtained the agreement to participate in this study from the head of the PHC.
2. The PI will ask the coordinator midwife at each PHC to introduce the names and phone numbers of the health cadres who will be potential participants. The PI and the researchers will contact each potential participant one by one to explain the procedure of this study and then obtain their consent to become a participant in this study. Cadres who belong to PHCs will receive the competency-based education program, and those who belong to PHCs allocated to the control group will follow the initial orientation provided by the PHC.
3. The PI and assistant (research team) will create a WhatsApp group for the intervention group and control group, and then distribute the questionnaires at an initial stage. All data will be collected at each PHC where the study will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Currently working as a health care for at least 1 year
2. Domiciled in the local area
3. Able to operate a telephone
4. Those who agreed to give consent and are willing to participate in the study
5. Those who agreed to receive the health education program and participate in the whole evaluation process.

Exclusion Criteria:

1. Those who are planning to move out to another city during the study period.
2. Those who are no longer work as a health cadre.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-02-17 (Actual)

PRIMARY OUTCOMES:
The competency level of health cadres | baseline (T0), after 1 month from the baseline (T1) and after 3 months from the baseline (T2)
  Competency is operationally defined as the ability to integrate components of knowledge, skills, values, and attitudes into practice, and build a trusting relationship with and guide a pregnant woman and her surroundings for them to take evidence-based appropriate behavior. The competency level is measured by the researcher developing a competency questionnaire which consists of a knowledge test, skill, and attitude checklist score

SECONDARY OUTCOMES:
The knowledge test scores of health cadres | baseline (T0), after 1 month from the baseline (T1) and after 3 months from the baseline (T2)
  researcher developing knowledge questionnaire
The health assessment skills checklist score of health cadres | after 1 month from the baseline (T1) and after 3 months from the baseline (T2)
  researcher developing health assessment skills checklist
The communication skills checklist score of health cadres | after 1 month from the baseline (T1) and after 3 months from the baseline (T2)
  researcher developing communication skills checklist
The confidence score of health cadres | after 1 month from the baseline (T1) and after 3 months from the baseline (T2)
  researcher developing communication skills checklist
The satisfaction score of health cadres | after 1 month from the baseline (T1)
  researcher developing satisfaction skills checklist

CONTACTS AND LOCATIONS:
Overall Officials: Dewie Sulistyorini, Principal Investigator — Hiroshima University
Locations (1):
- Politeknik Banjarnegara, Banjarnegara, Cental Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Share according to request to the PI and researcher
Time Frame: April 2025 - April 2026
Access Criteria: dewiesulistyorini@gmail.com

REFERENCES:
- [Derived] Sulistyorini D, Huq KATME, Babaita AO, Aivey SA, Huiying G, Kazawa K, Fukushima Y, Kako M, Moriyama M. Effectiveness of education programme to increase competency of health cadres in Indonesia: a cluster non-randomised controlled trial. BMJ Open. 2025 Dec 29;15(12):e095428. doi: 10.1136/bmjopen-2024-095428. PMID 41469067